CLINICAL TRIAL: NCT01881386
Title: Investigation of Lactate Measured Using Magnetic Resonance Spectroscopy as a Biomarker of Tumour Response
Brief Title: Lactate Imaging as a Tumour Biomarker
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: 13/LO/0536 CCR3939
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: Magnetic Resonance Spectroscopy; Lactate
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lymphoma: Lymphoma patients before and after receiving standard CHOP therapy
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- Metastatic Colorectal: Patients with metastatic colorectal cancer
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- Phase 1: Patients enrolled in Phase 1 clinical trials of new agents, whose mechanism of action is expected to lead to changes in lactate concentration
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- Brain: Patients with primary brain tumours and patients with cerebral lymphoma

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Spectroscopy
  Groups: Lymphoma; Metastatic Colorectal; Phase 1

SUMMARY:
This project is designed to investigate whether measurements of lactate in tumours, made using a magnetic resonance technique similar to MRI, is an effective non-invasive method to detect whether some new targeted drugs are having their desired effect.

The study hypothesis is that by using magnetic resonance spectroscopy techniques, we will be able to observe changes in tumour lactate levels in vivo, in response to treatment.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:lymphoma patients

* minimum lesion size of 2cm
* not pretreated but scheduled to be treated with CHOP (Cyclophosphamide, Hydroxydaunomycin,Oncovin and Prednisolone)

Cohort 2:Colorectal patients

* metastatic disease of at least 2cm
* not pretreated

Cohort 3:Phase 1 Drug Development

* minimum lesion size at least 2cm

Cohort 4: Brain

* primary brain tumours receiving radiotherapy and temozolomide
* cerebral lymphoma receiving standard chemotherapy

Exclusion Criteria:

* MRI incompatible metal implants
* Claustrophobia
* Inability to tolerate a 40 minute MRI scan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in MRS lactate measurements at two time points after treatment and clinical response | 7 and 21 days post treatment

SECONDARY OUTCOMES:
Reproducibility of MRS lactate measurement | Two baseline measurements taken at day -7 to 0 pre-treatment

OTHER OUTCOMES:
Correlation between changes in post treatment MRS lactate measurements and serum lactate dehydrogenase | Baseline and 7 and 21 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — ICR
Locations (1):
- The Institute of Cancer Research and Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom